CLINICAL TRIAL: NCT01186354
Title: Implications of Health and Genetic Literacy for Genomic Medicine
Brief Title: Understanding of Genetic Risk Information for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00021370; 1R21HL096573-01A1 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-08-23 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; health literacy; genetic literacy; genetic risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Receiving results via web-based program (Experimental): participants will receive genetic risk results for Type 2 diabetes via a web-based program that they access on their own
  Interventions: Behavioral: Receiving results via genetic counselor

INTERVENTIONS:
Behavioral: Receiving results via genetic counselor — participants will receive genetic risk information for Type 2 diabetes from a board certified genetic counselor
  Other Names: genetic counseling

SUMMARY:
This research study is being conducted to learn about how health and genetic literacy (i.e., how well a person understands health and genetic information) affects a person's ability to understand genetic risk information for Type 2 diabetes and whether that person chooses to change their lifestyle and health behaviors to reduce their risk. The investigators also want to learn if the manner in which the genetic risk information is communicated affects the level of understanding and potential behavior changes. Participants will be tested for genetic risk of developing Type 2 diabetes and will received results either via a web-based computer program, or in-person from a genetic counselor.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Speak fluent English
* Have an email address and access to the internet
* Not diagnosed with type 2 diabetes

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Accurate understanding of genetic risk information | assessed at follow-up 1 week, 3 months and 6 months after receiving results

SECONDARY OUTCOMES:
Impact on behavior change | assessed upon follow-up (3 mon, 6 mon)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne B Haga, PhD, Principal Investigator — Duke University Medical Center, Institute for Genome Sciences and Policy
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Mills R, Powell J, Barry W, Haga SB. Information-seeking and sharing behavior following genomic testing for diabetes risk. J Genet Couns. 2015 Feb;24(1):58-66. doi: 10.1007/s10897-014-9736-1. Epub 2014 Jun 14. PMID 24927802
- [Derived] Haga SB, Barry WT, Mills R, Svetkey L, Suchindran S, Willard HF, Ginsburg GS. Impact of delivery models on understanding genomic risk for type 2 diabetes. Public Health Genomics. 2014;17(2):95-104. doi: 10.1159/000358413. Epub 2014 Feb 27. PMID 24577154
- [Derived] Haga SB, Barry WT, Mills R, Ginsburg GS, Svetkey L, Sullivan J, Willard HF. Public knowledge of and attitudes toward genetics and genetic testing. Genet Test Mol Biomarkers. 2013 Apr;17(4):327-35. doi: 10.1089/gtmb.2012.0350. Epub 2013 Feb 13. PMID 23406207
- [Derived] Waxler JL, O'Brien KE, Delahanty LM, Meigs JB, Florez JC, Park ER, Pober BR, Grant RW. Genetic counseling as a tool for type 2 diabetes prevention: a genetic counseling framework for common polygenetic disorders. J Genet Couns. 2012 Oct;21(5):684-91. doi: 10.1007/s10897-012-9486-x. PMID 22302620